CLINICAL TRIAL: NCT02485236
Title: Randomized Nasal High Flow Therapy Versus Oxygen Supplementation in Postoperative Care of Obstructive Sleep Apnea Patients With Continuous Positive Airway Pressure Non-Compliance
Brief Title: Postoperative Nasal High Flow Versus Oxygen for Positive Airway Pressure Non-Compliance Sleep Apnea Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bernardo J. Selim, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-000716
Record Dates: First submitted 2015-06-09; First posted 2015-06-30 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low flow oxygen via nasal cannula (Active Comparator): In the low flow oxygen via nasal cannula, patients will be supplemented with 1 liter per minute via nasal cannula. Adjustment of initial setting upon floor arrival: To adjust oxygen 1-4 liters per minute to an arterial oxygen saturation of > 88%. Continuous oximetry will be collected up to 48 hours. Standard postsurgical care.
  Interventions: Device: Low flow oxygen via nasal cannula
- Humidified Nasal High Flow Therapy (Active Comparator): Adjustment of humidified high flow air therapy: To adjust oxygen 1-4 liters per minute to an arterial oxygen saturation of > 88%. To adjust air flow to patient comfort (20-35 liters per minute). Continuous oximetry will be collected up to 48 hours. Standard postsurgical care.
  Interventions: Device: Humidified Nasal High Flow Therapy

INTERVENTIONS:
Device: Low flow oxygen via nasal cannula — In the low flow oxygen group, patients will be supplemented with 1 liter per minute via nasal cannula. Adjustment of initial setting upon floor arrival: To adjust oxygen 1-4 liters per minute to an arterial saturation of oxygen of > 88%. Continuous oximetry will be collected up to 48 hours. Standard postsurgical care.
  Arms: Low flow oxygen via nasal cannula
Device: Humidified Nasal High Flow Therapy — Adjustment of initial setting upon floor arrival: To adjust oxygen 1-4 liters per minute to arterial saturation of oxygen > 88%. To adjust air flow to patient comfort (20-35 liters per minute). Continuous oximetry will be collected up to 48 hours. Standard postsurgical care.
  Other Names: Airvo 2 from Fisher and Paykel
  Arms: Humidified Nasal High Flow Therapy

SUMMARY:
The study aims to compare the efficacy of Nasal High Flow Therapy (NHF) with low-flow oxygen supplementation in improving postoperative intermittent desaturations. If so, this mode of therapy would provide a cost effective, relatively easy to implement, and better tolerated treatment to Continuous Positive Airway Pressure (CPAP) for oxygen stabilization.

DETAILED DESCRIPTION:
Patients identified preoperatively with previously diagnosed obstructive sleep apnea (intermittent collapse of upper airway while asleep) who refuse Continuous Positive Airway Pressure use after surgery and are treated with routine postoperative supplemental oxygen alone (1 liters per minute) will have more oscillation of oxygen saturation during the night (measure by overnight oximetry) than those treated with high nasal flow air insufflator (Fisher & Paykel Airvo 2 device) with same amount of oxygen supplement (1 liters per minute).

ELIGIBILITY:
Inclusion Criteria:

1. Known diagnosis of obstructive sleep apnea by polysomnography (Apnea Hypopnea Index ≥ 5 events per hour) with recommendation of Continuous Positive Airway Pressure use.
2. The patient declines use of Continuous Positive Airway Pressure for the upcoming elective surgery.
3. The patient will require more than 48 hours of hospitalization.
4. Informed consent obtained from patient or approved designate.

Exclusion Criteria:

1. Predetermined need for Continuous Positive Airway Pressure post-operatively by surgical team.
2. Body Mass Index ≥ 40.
3. Patient with congestive heart failure and diagnosis of Cheyne- Stokes respiration or central apnea.
4. Patients who are oxygen dependent due to moderate to severe Chronic Obstructive Pulmonary Disease (Available Forced Expiratory Volume at 1 second of < 50% predicted) or advanced interstitial lung disease.
5. Preexisting chronic hypercapnia with known neuromuscular disease with respiratory involvement (e.g. Amyotrophic Lateral Sclerosis, myopathy).
6. Severe anemia necessitating blood transfusion.
7. Presence of tracheostomy.
8. Naso-oral malformation or severe nasal septal defect.
9. Presence of dementia or other diagnosed neurodegenerative disease.
10. Non-English speakers
11. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-05-28 (Actual); Study Completion 2017-05-28 (Actual)

PRIMARY OUTCOMES:
The 4% change oxygen-desaturation index (4% ODI) determined by pulse oximetry | At 48 hours postsurgery
  The 4% change oxygen-desaturation index (4% ODI) as determined from the recorded pulse oximetry data during the first postoperative 48 hours.

SECONDARY OUTCOMES:
Incidence rate of postoperative cardio-respiratory complications | At 48 hours postsurgery
  Incidence rate of postoperative cardio-respiratory complications such as Intensive Care Unit transfer, acute arrhythmia, myocardial ischemic event, delirium, new infiltrate or atelectasis, and any complication (combination of two or more of those above)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo J. Selim, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials